CLINICAL TRIAL: NCT04726943
Title: Radiofrequency Energy Applications Targeting Significant Residual Leaks After Left Atrial Appendage Occlusion
Brief Title: RF Applications for Residual LAA Leaks
Acronym: REACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCAI_RFLK01
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Left Atrial Appendage Thrombosis; Stroke, Ischemic; Atrial Fibrillation
Keywords: stroke; atrial fibrillation; left atrial appendage; prevention; leak; radiofrequency
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RF Energy (Experimental): RF delivery targeting the atrial side of a significant residual leak in patients with acute and chronic evidence of incomplete percutaneous LAA occlusion
  Interventions: Procedure: Radiofrequency Energy Applications

INTERVENTIONS:
Procedure: Radiofrequency Energy Applications — RF energy applications to the atrial edge of a leak resulting from incomplete LAA occlusion

SUMMARY:
Although the clinical impact of residual left atrial appendage (LAA) leaks still requires confirmation, its patency resulting from incomplete LAA closure may promote blood stagnation and thrombus formation, and increase the risk of thromboembolic events. The main purpose of this trial is to evaluate the safety and efficacy of percutaneous leak closure with radiofrequency energy applications.

DETAILED DESCRIPTION:
Therapies locally targeting the LAA via occlusion, exclusion, or excision have emerged as an alternative and effective approach for stroke prophylaxis in AF patients, especially those with OAC contra-indications. Despite mounting evidence of their safety and efficacy in comparison with standard oral therapy, device-related thrombus and incomplete LAA closure resulting in residual, significant leak may occur, potentially hindering an effective stroke prevention. Radiofrequency energy has been adopted in several settings (e.g., vascular, orthopedic, aesthetic surgery) to achieve thermal-induced tissue retraction.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years.
2. Presence of a significant LAA leak acutely or at follow-up.
3. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Life expectancy < 2 years.
2. pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
3. presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | 1-3 months
  Complete LAA occlusion or presence of a mild/minimal peri-device leak on FU TEE

SECONDARY OUTCOMES:
Peri-Procedural Success | Peri-Procedural
  Complete LAA occlusion or presence of mild/minimal (1-2 mm) residual leak assessed via multiplane color Doppler imaging on TEE/ICE at the end of the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - St. David's Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Della Rocca DG, Murtaza G, Di Biase L, Akella K, Krishnan SC, Magnocavallo M, Mohanty S, Gianni C, Trivedi C, Lavalle C, Forleo GB, Natale VN, Tarantino N, Romero J, Gopinathannair R, Patel PJ, Bassiouny M, Del Prete A, Al-Ahmad A, Burkhardt JD, Gallinghouse GJ, Sanchez JE, Doshi SK, Horton RP, Lakkireddy D, Natale A. Radiofrequency Energy Applications Targeting Significant Residual Leaks After Watchman Implantation: A Prospective, Multicenter Experience. JACC Clin Electrophysiol. 2021 Dec;7(12):1573-1584. doi: 10.1016/j.jacep.2021.06.002. Epub 2021 Jul 27. PMID 34330671